CLINICAL TRIAL: NCT00983567
Title: An Interactive Web-Based Program to Improve Food and Activity Choices of Teens
Acronym: Teen Web
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Karen Cullen, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2007-55215-17998; USDA 2007-55215-17998
Record Dates: First submitted 2009-07-30; First posted 2009-09-24 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Diet; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Teen web (Experimental): Main web - with all components
  Interventions: Other: teen web
- Minimal teen web (Active Comparator): Teen web minus behavioral components
  Interventions: Other: teen web

INTERVENTIONS:
Other: teen web — Min web

SUMMARY:
This study will test a website for teens designed to help them improve both diet and physical activity. The website will have several components: educational messages, role model stories, goal setting, self-monitoring forms, problem solving, a monitored discussion forum, and diet and physical activity (PA) assessment questionnaires.

DETAILED DESCRIPTION:
Increasing numbers of youth are at risk for becoming overweight because of poor diets and low physical activity levels. Prevention is key to reducing the obesity problem. Intervention programs must be easily accessible, and include intervention materials in a format that draws attention and interest. This study evaluates an 8-week web-based intervention for teens to promote healthy food and physical activity choices. The web program includes role model stories, nutrition and activity information pieces, goal setting and problem solving, and self-monitoring. Students will complete assessments at baseline, 8-weeks post, and then 6 and 12-months post intervention.

ELIGIBILITY:
Inclusion Criteria:

* ability to speak English
* 12-17 years old

Exclusion Criteria:

* no special diets

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2009-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
diet (fruit, vegetables, sweetened beverages, fat) | baseline, post, 6-and 12-months

SECONDARY OUTCOMES:
BMI | baseline, post, 6- and 12-months
Physical activity:self-report | baseline, post, 6-and 12-months

CONTACTS AND LOCATIONS:
Overall Officials: Karen W Cullen, DrPH, Principal Investigator — Baylor College of Medicine
Locations (1):
- Children's Nutrition Research Center, Houston, Texas, United States